CLINICAL TRIAL: NCT03071003
Title: A Randomised Double Blind, Multiple Dose, Pharmacokinetic and Safety Study of SENS 401 in Healthy Subjects
Brief Title: A Study of SENS 401 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Simbec Research (Industry)
Collaborators: Sensorion (Industry)
Responsible Party: Principal Investigator, Robert Adams, Prinicipal Investigator, MBBS, Simbec Research
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: RD716/33196
Record Dates: First submitted 2017-02-22; First posted 2017-03-06 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Inner Ear Disease
Keywords: Pharmacokinetics; Healthy Volunteer Study
MeSH Terms: conditions — Labyrinth Diseases | interventions — SENS-401

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 SENS 401 & Placebo (Experimental): 12 subjects will receive 29 mg SENS-401 (approximately 4 male and 4 female subjects) or placebo (approximately 2 male and 2 female subjects) once daily for 7 days.
  Interventions: Drug: SENS-401; Drug: Placebo
- Cohort 2 SENS 401 & Placebo (Experimental): 12 subjects will receive 29 mg SENS-401 (approximately 4 male and 4 female subjects) or placebo (approximately 2 male and 2 female subjects) twice daily for 6 days and a single dose of 29 mg SENS-401 or placebo in the morning on Day 7.
  Interventions: Drug: SENS-401; Drug: Placebo
- Cohort 3 SENS 401 & Placebo (Experimental): 12 subjects will receive 43.5 mg SENS-401 (approximately 4 male and 4 female subjects) or placebo (approximately 2 male and 2 female subjects) twice daily for 6 days and a single dose of 43.5 mg SENS-401 or placebo in the morning on Day 7.
  Interventions: Drug: SENS-401; Drug: Placebo

INTERVENTIONS:
Drug: SENS-401 — Oral Administration
Drug: Placebo — Oral Administration

SUMMARY:
Sensorion are the study sponsor and the objective of this study is to investigate the safety and pharmacokinetic (PK) profile of SENS 401 in humans after a single and repeat dose administration and to confirm that, there is no interconversion of the (R) enantiomer to the (S) enantiomer.

The study only involves the one drug, referred to as SENS-401.The key objective is to assess the safety of SENS 401 after multiple doses in healthy subjects.

The population who are eligible to take part in the study are healthy male and female, non-smoking volunteers, aged between 18 and 50 years, as determined by screening tests at Simbec.

Participation in the trial will last for about 3 weeks (from first screening to final end of study visit).

DETAILED DESCRIPTION:
This is a randomised, double blind, multiple dose, safety and PK study. Three cohorts of 12 subjects will be administered with three different dose regimens.

Screening assessments will be carried out within 14 days before administration of the investigational medicinal product (IMP). Eligible subjects will be asked to return for the treatment period.

Cohort 1: 12 subjects will receive 29 mg SENS-401 or placebo once daily for 7 days.

Cohort 2: 12 subjects will receive 29 mg SENS-401 or placebo twice daily for 6 days and a single dose of 29 mg SENS-401 or placebo in the morning on Day 7.

Cohort 3: 12 subjects will receive 43.5 mg SENS-401 or placebo twice daily for 6 days and a single dose of 43.5 mg SENS-401 or placebo in the morning on Day 7.

Subjects will be asked to attend Simbec 5-7 days after administration of the last dose for a post study visit. If they are withdrawn from the study, they will still be asked to attend for an end of study assessment. Subjects may be asked to return again if we need to follow them up.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females (non pregnant/non lactating) between 18 and 50 years of age.
2. Female subject of child bearing potential with a negative pregnancy test at the screening visit and willing to use 2 effective methods of contraception, from first dose until 3 months afterwards (i.e., until 3 months after last SENS-401 dose).
3. Female subject of non child bearing potential with negative pregnancy test at the screening visit. For the purposes of this study, this is defined as the subject being amenorrheic for at least 12 consecutive months or at least 4 months post surgical sterilisation (including bilateral fallopian tube ligation or bilateral oophorectomy with or without hysterectomy) and levels of follicle stimulating hormone (FSH) falling within the respective pathology reference range. In the event a subject's menopause status has been clearly established (for example, the subject indicates she has been amenorrheic for 10 years), but FSH levels are not consistent with a post menopausal condition, determination of subject eligibility will be at the discretion of the Investigator following consultation with the Sponsor's Responsible Physician.
4. Male subject willing to use 2 effective methods of contraception, (unless anatomically sterile) from first dose until 3 months afterwards (i.e., until 3 months after last SENS-401 dose).
5. Subject with a body mass index (BMI) of 18 30 kg/m2. If Asians are included, BMI values will be modified to 16-23 kg/m2 (this range is considered as normal in Asian population). BMI = body weight (kg)/height (m)2.
6. Subject with no clinically significant abnormal serum biochemistry, haematology and urine examination values within 14 days of the first dose.
7. Subject with a negative urinary drugs of abuse screen, determined within 14 days of the first dose (a positive alcohol result may be repeated at the discretion of the Investigator).
8. Subject with negative human immunodeficiency virus (HIV), hepatitis B surface antigen (Hep B) and hepatitis C virus antibody (Hep C) results.
9. Subject with no clinically significant abnormalities in 12 lead electrocardiogram (ECG) determined within 14 days of the first dose.
10. Subject with no clinically significant abnormalities in blood pressure or pulse determined within 14 days of the first dose.
11. Subject is a non smoker or ex smoker who has not smoked in the last 3 months (determined by urine cotinine < 500 ng/mL at screening visit).
12. Subject is available to complete the study (including all follow up visits) and comply with study restrictions.
13. Subject satisfies a medical examiner about their fitness to participate in the study.
14. Subject provides written informed consent to participate in the study.

Exclusion Criteria:

1. Subject with a clinically significant history of gastrointestinal disorder likely to influence drug absorption.
2. Subject in receipt of regular medication (with the exception of contraception) within 14 days of the first dose that may have an impact on the safety and objectives of the study (Investigator's discretion).
3. Subject with evidence of renal, hepatic, central nervous system, respiratory, cardiovascular or metabolic dysfunction.
4. Subject with any renal (serum creatinine (CREAT) level > 1.5 fold above the upper limit of normal (ULN) or liver insufficiency (alkaline phosphatase (ALP) level > 1.2 fold above ULN, gamma glutamyl transferase (GGT), aspartate transaminase (AST), or alanine transaminase (ALT) level > 2.5 fold above ULN, and total bilirubin (BIL T) level > 1.5 fold above ULN).
5. Subject with history of, or family history (immediate relative) of, long QT syndrome or Torsade de Pointes or symptomatic bradycardia.
6. Subject with clinically significant history of previous allergy / sensitivity to SENS-218 or its excipients or other 5-hydroxytryptamine (5 HT3) receptor antagonists.
7. Subject with a clinically significant history of drug or alcohol abuse.
8. Subject with inability to communicate well with the Investigator (i.e., language problem, poor mental development or impaired cerebral function).
9. Subject participation in a New Chemical Entity clinical study within the previous 4 months or a marketed drug clinical study within the previous 3 months. (N.B. washout period between studies is defined as the period of time elapsed between the last dose of the previous study and the first dose of the next study).
10. Subject donated 450 mL or more blood within the previous 3 months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-10-21 (Actual); Primary Completion 2017-03-21 (Actual); Study Completion 2017-10-16 (Actual)

PRIMARY OUTCOMES:
Safety of SENS 401 after multiple doses in healthy subjects | Throughout the study until post study visit (A period of approximately 4 weeks)
  AEs

SECONDARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | Day 1-9
  Cohort 1, 2 and 3 - Day 1 and Day 7 Cmax
Area under the curve 0 to 24 [AUC0-24] | Day 1-9
  Cohort 1 [AUC0-12], Cohort 2 and 3 [AUC0-24]
Interconversion of the (R) enantiomer (SENS-401) and (S)-enantiomer (SENS-219) in human plasma. | Day 1-9
  Individual SENS-401,SENS-219 and SENS-218 concentration-time data following administration of SENS-401 will be listed.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Adams, MBBS, Principal Investigator — Simbec Research
Locations (1):
- Simbec Research, Merthyr Tydfil, United Kingdom

IPD SHARING:
Plan to Share IPD: No